CLINICAL TRIAL: NCT03999242
Title: Clinical Significance of Charcot-Leyden Crystals in Bronchial and Sinonasal Pathological Samples
Brief Title: Charcot Leyden Crystals in Pathology
Acronym: CLCpath
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0256
Record Dates: First submitted 2019-05-20; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: nasal polyposis; rhinosinusitis; Charcot Leyden Crystals; Eosinophils
MeSH Terms: conditions — Asthma; Nasal Polyps; Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Bronchial biopsies, sinonasal biopsies, BAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Charcot Leyden crystals (CLC) are sometime reported in pathological reports of airway or sinonasal samples but their clinical significance remain elusive. The investigators organized a retrospective analysis of all consecutive patients with CLC seen at our institution between 1986 and 2019

DETAILED DESCRIPTION:
In recent years, improved knowledge of eosinophilic inflammation has led to the approval of biologics aimed at inhibiting the pathways of eosinophilic activation, notably via the interleukin 5 pathway in eosinophilic asthmatic patients uncontrolled despite receiving maximum doses of standard drugs. These treatments showed efficacy in asthmatic patients with a high level of eosinophils in their induced sputum (> 3%) and the criteria were extended to those with circulating eosinophilia (> 300 / mm3). Eosinophils are therefore an important biomarker for phenotyping asthmatic patients. The Charcot-Leyden crystals are a reflection of the presence of eosinophils, and are sometimes found in some pathological samples. It is hypothesized that the presence of Charcot-Leyden crystals, a reflection of tissue eosinophilia, is a predictive factor for the efficacy of anti-IL5 biotherapies in patients with severe eosinophilic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Having Charcot Leyden Crystals in a pathological sample

Exclusion Criteria:

* Having Charcot Leyden Crystals in a pathological sample taken outside the airways the nose and the sinus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients seen at our institution
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
'Level of asthma control/severity according to GINA stepwise approach | Baseline (day 0)
'Level of asthma control/severity according to GINA stepwise approach | Baseline (day 0) to Month 12

SECONDARY OUTCOMES:
Cumulative annualized dose of inhaled and systemic corticosteroids | Baseline (day 0) to Month 12
  The quantity of corticosteroids consumed during the course of a year.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Bourdin, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC